CLINICAL TRIAL: NCT01799369
Title: Surgical Apgar Score in Clinical Practice: a Pilot Study
Acronym: SAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Surgical Research Group (Other)
Collaborators: National Health Service, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: LSRG-001
Record Dates: First submitted 2013-02-23; First posted 2013-02-26 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Postoperative Care
Keywords: Surgical Apgar Score

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Routine post-operative care
- Intervention (Experimental): Post-operative care influenced by the Surgical Apgar Score
  Interventions: Behavioral: Surgical Apgar Score

INTERVENTIONS:
Behavioral: Surgical Apgar Score — Post-operative care influenced by Surgical Apgar Score
  Arms: Intervention

SUMMARY:
Background Surgeons lack a routine, objective evaluation of patient condition after surgery. We currently rely on subjective assessment of available patient data. The current scoring methods such as Acute Physiology and Chronic Health Evaluation and Physiological and Operative Severity Score for the enUmeration of Mortality and morbidity are complex and cumbersome and have therefore not been adopted into routine practice.

The Surgical Apgar Score (SAS) is a simple score on a scale of 0 to 10 calculated from 3 parameters collected during the operation: lowest heart rate, lowest blood pressure, estimated blood loss (Regenbogen et al., Arch Surg 2009).

Previous validation studies have shown a good correlation between the score and incidence of major complications or death occurring within 30 days. For example, 75% patients with a score of 0-2 had major complications, whereas it was only 5% in those with a score of 9-10. To date, the SAS has never been clinically applied and tested in a trial.

We believe that routine use of the SAS will lead to a reduction in major complications and deaths after surgery. We also believe that it will lead to a reduction in the severity of the complications.

This is based on our theory that the SAS eliminates the guesswork. Using this score will add objectivity and clarity to clinical decisions that are presently based on clinical instinct or 'gut feeling'. The score will more clearly highlight those patients who are at an increased risk of developing complications or dying and will flag them up for increased monitoring, a higher index of clinical suspicion and a lower threshold for early management of problems.

Primary Aim The primary aim of the pilot is to strengthen the design and assess the feasibility of the main study on the SAS. We aim to recruit 100 patients in each group, 200 in total. The primary aim of the main study will be to establish if clinical application of the SAS leads to a reduction in 30-day post-operative morbidity and mortality.

Study Design The design of this pilot is the same as what the main trial will eventually be: a multicentre single-blind randomised controlled trial (RCT). Current data suggests the overall expected major complication or death rate in our target population would be 21%. The sample size of the future RCT is therefore estimated to be 986 each group to detect a 5% reduction in complications (Significance 0.05%, Power 80%).

Outcomes Our primary outcome will be major complications or death within 30 days of operation. Our secondary outcomes (all within 30 days of operation) will be minor complications, primary and secondary critical care admissions and length of stay, duration of therapeutic antibiotics, number of additional operations under general anaesthetic to treat complications, and overall length of stay.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18y+)
* General or vascular surgery
* Elective or emergency surgery
* Routine outpatient follow-up required

Exclusion Criteria:

* Those without capacity to consent to involvement in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2011-04; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Major complications or death | 30 days
  Composite binary outcome

CONTACTS AND LOCATIONS:
Overall Officials: James B Haddow, MRCS, Study Chair — London Surgical Research Group

REFERENCES:
- [Result] Haddow JB, Adwan H, Clark SE, Tayeh S, Antonowicz SS, Jayia P, Chicken DW, Wiggins T, Davenport R, Kaptanis S, Fakhry M, Knowles CH, Elmetwally AS, Geddoa E, Nair MS, Naeem I, Adegbola S, Muirhead LJ; London Surgical Research Group. Use of the surgical Apgar score to guide postoperative care. Ann R Coll Surg Engl. 2014 Jul;96(5):352-8. doi: 10.1308/003588414X13946184900840. PMID 24992418